CLINICAL TRIAL: NCT03761147
Title: Women's First Gastrointestinal Activation Post-elective Cesarean Birth During Post-partum Hospitalization:A Comparison of Paula Method (the Circular Exercises Method) to Standard Care
Brief Title: Gastrointestinal Activation Post-elective CS (Cesarean Section) :A Comparison of Paula Method to Standard Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI PAULA-HMO-CTIL
Record Dates: First submitted 2017-11-26; First posted 2018-12-03 (Actual); Results first posted 2021-08-12 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2020-05

CONDITIONS: Bowel Dysfunction
MeSH Terms: conditions — Intestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paula Method (Experimental)
  Interventions: Other: Paula exercises
- Standard of Care (No Intervention)

INTERVENTIONS:
Other: Paula exercises — structured exercises aimed to stimulate ring muscles
  Arms: Paula Method

SUMMARY:
Women generally report discomfort and a delay in GI motility after CS. The Paula method, circular exercises of ring muscles has been shown to increase GI motility. This method had not been studied in women post CS. The current study is comparing the resumption of bowel sounds after CS in women utilizing the Paula exercises to standard care (no exercises).

ELIGIBILITY:
Inclusion Criteria:

* Elective, singleton, term CS, with spinal or epidural anesthesia

Exclusion Criteria:

* GI/ absorption disorders (Chron's, IBS)
* general anesthesia
* urgent CS

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liebergall-Wischnitzer M, Shaphir A, Solnica A, Hochner-Celnikier D. Are Paula method exercises effective for gastrointestinal reactivation post-elective cesarean delivery? Randomized controlled trial. J Adv Nurs. 2021 Apr;77(4):2026-2032. doi: 10.1111/jan.14681. Epub 2020 Nov 29. PMID 33249611

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard of Care: Standard of Care
Period: Overall Study
Arm/Group | Paula Method | Standard of Care
Started | 32 | 32
Completed | 25 | 28
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paula Method | Standard of Care | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.65 (6.32) | 34.62 (5.15) | 35.14 (5.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 64
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 32 | 32 | 64
Region of Enrollment [Number; unit: participants]
  Israel | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Time to the Resumption of Bowel Functioning as Assessed by Flatus Passage
Description: flatus passage
Time Frame: 72 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Paula Method | Standard of Care
Number analyzed (Participants) | 25 | 28
hours | 24.1 (6.85) | 39.1 (10.4)
Statistical Analysis 1: Comparison: Paula Method vs Standard of Care; Test type: Superiority; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 96 hours
Arm/Group | Paula Method | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT03761147/Prot_SAP_000.pdf